CLINICAL TRIAL: NCT05463562
Title: Detection of Multimodal Biomarkers of Electroconvulsive Therapie in Severe and Treatment-resistent Depression
Brief Title: Multimodal Biomarkers of Electroconvulsive Therapy in Severe and Treatment-resistant Depression
Acronym: DetECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Other Study IDs: 21-1087
Record Dates: First submitted 2022-07-11; First posted 2022-07-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Depressive Disorder; Bipolar Disorder
Keywords: electroconvulsive therapy; biomarkers; genetics; depression; prediction; molecular neuroscience
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Electroconvulsive therapy (ECT) is a widespread and safe stimulation method that has been used successfully for decades in psychiatric diseases such as severe or therapy-resistant depression. Unfortunately, ECT still has stigmas attached to it. The latter often leads to reservations among those affected and perturbs optimal and guideline-based therapy. Despite the demonstrated effectiveness of ECT, prediction of treatment response is still not possible. This is due to the limited knowledge about the biological mechanisms of action of ECT, especially on an individuum level. Thus, the DetECT study intends to recruit 134 inpatient subjects of the Max Planck Institute of Psychiatry with severe and/or treatment resistant depression receiving ECT to perform weekly psychometry and blood draws before and after ECT sessions one, seven, and twelve. The subsequent biopsychological analysis comprises omics, physiological, neurocognitive, and psychometric measurements. The multimodal data collected will be used to identify data-driven clusters associated with ECT mechanisms and outcome.

DETAILED DESCRIPTION:
Background:

With around 320 million cases, depression is one of the most common psychiatric disorders worldwide. In addition to psychopharmacological treatment and psychotherapy, ECT is a common treatment option. This technique is referred to as the gold standard of stimulation procedures due to its good effectiveness and safe application. Despite the widespread use of ECT, knowledge of the underlying biological processes that lead to symptom improvement is still limited. Accordingly, there are no clinical-psychological or biological biomarkers that can reliably predict the course of the disease or the response to ECT in individual cases. Due these circumstances, the primary aim of the present DetECT study is to identify individual parameters or clusters of biological and psychological-clinical features that are associated with the course of depression under ECT.

Material and Methods:

The monocentric, explorative-prospective DetECT study (planned total duration: 3 years) recruits adult and legally competent patients who receive inpatient treatment at the Max Planck Institute for Psychiatry and undergo ECT for a severe depressive episode. Participants will have a total of five (in select cases: seven) venous blood samples taken over an average of seven weeks, that is parallel to the first twelve ECT session on three treatment days (total volume: ~124 ml; in select cases 152 ml). All participants will also be asked to complete self-rating questionnaires on their depressive and neurocognitive symptoms (Patient Health Questionnaire 9 and 15, Questionnaire on Mental Capacity, Beck Depression Inventory II) each week. At the beginning, in the middle and at the end of the seven-week study period, three external assessment questionnaires (Montgomery-Åsberg Depression Rating Scale, Hamilton Rating Scale for Depression, Global Assessment of Functioning) are collected by the study staff. In addition, medical, anamnestic and sociodemographic information on the course of illness and therapy is extracted from the patient records. All biomaterials and data collected in the DetECT study, together with the samples and data from the Max Planck of Psychiatry's biobanking, are double pseudonymised or anonymised and stored for 10 or 30 years, depending on subject preference. Protecting the privacy and rights of the study participants is our top priority. All analyses are performed only by using the participant's study code to guarantee a maximum of data security. Modern and multidimensional analysis techniques will be employed to the biopsychological parameters and to the clinical and socioeconomic information. On a group or subgroup level, this will likely help to link multidimensional biomarker clusters with treatment outcome under ECT.

Discussion:

Taken together, the DetECT study aims to improve the quality of psychiatric treatment of severely depressed patients. The investigators argue that the study novelty lies in its longitudinal and multimodal data collection and analysis approach. This could effectively advance personalization and specification of ECT indication and application. Ultimately as well as in a nutshell, the overall study objective is to identify those patients who benefit most from in terms of the effect/side-effect profile.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (of legal age, legally competent) and desire to participate
* Diagnosis of a depressive episode (also in the case of bipolar affective disorder) or depression according to the ICD-10 or ICD-11 or DSM-4 or DSM-5
* Indication and planned electroconvulsive therapy
* Signed Electroconvulsive Therapy Informed Consent Form
* Consent to participate by personally signing the declaration of consent including data protection concept and data use for the DetECT study
* Consent and participation in MPI of Psychiatry's biobanking

Exclusion Criteria:

* Age < 18 years (minor)
* Pregnancy and breastfeeding
* Existence of legal supervision
* Pervasive developmental disorders and/or intellectual disability
* Acute, relevant substance abuse of alcohol, over-the-counter and prescription drugs, or illicit drugs
* Severe neurological disease (especially severe organic brain damage)
* Acute, serious general illness (especially clinically relevant, aplastic and/or anemia requiring transfusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only persons of legal age who are in inpatient psychiatric treatment at the Max Planck Institute for Psychiatry and have given consent to participate in local biobanking can take part in the present DetECT study.
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-02-23 (Estimated); Study Completion 2025-02-23 (Estimated)

PRIMARY OUTCOMES:
Genetics | baseline
  Genotyping based on material extracted from peripheral blood
Changes in gene expression over time | baseline, week 4, week 7
  Longitudinal analysis of mRNA extracted from peripheral blood
Changes in epigenetics including gene methylation and miRNA expression over time | baseline, week 4, week 7
  Longitudinal analysis of DNA methylation and miRNA expression from peripheral blood
Protein, lipid, and electrolyte changes over time | baseline, week 4, week 7
  Longitudinal analysis of blood-based proteins (e.g. CRP, IL6), lipids (e.g. cholesterol), electrolytes, and other molecules from peripheral blood
Changes in immunophenotyping over time | baseline, week 4, week 7
  Longitudinal phenotyping of different immune cell populations from peripheral blood mononuclear cells (PBMCs)
Changes in purinergic signalling over time | baseline, week 4, week 7
  Longitudinal measurement of purines and pyrimidines as well as their metabolites in peripheral blood
Changes in body mass index (BMI) over time | baseline, week 4, week 7
  Longitudinal analysis of body mass index (BMI)
Changes in blood pressure over time | baseline, week 4, week 7
  Longitudinal analysis of blood pressure
Clinical and socioeconomic factors | baseline
  Influence on treatment response
Change from baseline in the Hamilton Depression Rating Scale (HAM-D) | Baseline, week 4, and week 7
  The HAM-D measures the presence and severity of depression. Each of the items is rated by a study clinician or trained study staff member and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the HAM-D score is ≤ 7 points
Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, week 4, and week 7
  The MADRS measures the presence and severity of depression. Each of the terms is rated by a study clinician or trained study staff member and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the MADRS score falls short of 12 points
Change from baseline in the Global Assessment of Functioning (GAF) | Baseline, week 4, and week 7
  The GAF approximates the level of symptom burden and psychosocial as well as occupational functioning in daily life. It is tailored primarily to psychiatric patients. It is rated from 0 to 100 by a trained clinician. The GAF score is a continuous variable and allows to estimate symptom reduction and functional assessment from a foreign rater perspective
Change from baseline in the Beck-Depression-Inventory II (BDI-II) | weekly
  The BDI-II measures the presence and severity of depression symptoms on a mostly psychological and partially somatic level. Each of the 21 items is rated by the patient and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the BDI-II score is ≤ 10 points
Change from baseline in the Patient Health Questionnaire 9 (PHQ-9) | weekly
  The PHQ-9 is a brief measure of depression symptoms. Each of the 9 items is rated by the patient from 0 = not at all to 3 = nearly every day and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the PHQ-9 score is ≤ 5 points.
Change from baseline in the Patient Health Questionnaire 15 (PHQ-15) | weekly
  The PHQ-15 is a measure of somatic symptom load in psychiatric disorders. Each of the 15 somatic symptoms is rated by the patient from 0 = not affected to 2 = strongly affected and added up to a summary score. Cut-off values are ≥ 5points (mild), ≥ 10 points (moderate), ≥ 15 points (severe) and represent somatization
Change from baseline in the Questionnaire on Mental Capacity (FLEI = dt. Fragebogen zur geistigen Leistungsfähigkeit) | weekly
  The FLEI measures neurocognitive functioning in the following domains: attention, memory, executive function, control scale. Each of the 35 questions is answered by the patient from 0 = never to 4 = very often. Summary scores are computed for the different neurocognitive domains. Since the FLEI is primarily a continuous variable, symptom reduction is commonly assessed quantitively

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Binder, MD, PhD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Mucke-Heim IA, Pape JC, Grandi NC, Erhardt A, Deussing JM, Binder EB. Multiomics and blood-based biomarkers of electroconvulsive therapy in severe and treatment-resistant depression: study protocol of the DetECT study. Eur Arch Psychiatry Clin Neurosci. 2024 Apr;274(3):673-684. doi: 10.1007/s00406-023-01647-1. Epub 2023 Aug 30. PMID 37644215